CLINICAL TRIAL: NCT01936948
Title: Safety of Endoscopic Resection of Large Colorectal Polyps: A Randomized Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Dartmouth College (Other); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Heiko Pohl, Principal Investigator, White River Junction Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPHS-23578
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Colon Polyps
Keywords: Large colon polyps; Polyp resection; Colon cancer screening; Colonoscopy; Endoscopic mucosal resection
MeSH Terms: conditions — Colonic Polyps | interventions — Surgical Instruments

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Clip closure + EndoCut (Active Comparator): Clipping of the mucosal defect after resection of a ≥20mm non-pedunculated study polyp using clips. Resection is done using the EndoCut electrocautery mode.
  Interventions: Procedure: Clip closure
- Clip closure + Coagulation (Active Comparator): Clipping of the mucosal defect after resection of a ≥20mm non-pedunculated study polyp using clips. Resection is done using the Coagulation electrocautery mode.
  Interventions: Procedure: Clip closure
- No clip closure + EndoCut (No Intervention): No clipping of the mucosal defect after resection of a ≥20mm non-pedunculated study polyp. Resection is done using the EndoCut electrocautery mode.
- No clip closure + Coagulation (No Intervention): No clipping of the mucosal defect after resection of a ≥20mm non-pedunculated study polyp. Resection is done using the Coagulation electrocautery mode.

INTERVENTIONS:
Procedure: Clip closure — Patients will be randomized to either closing the mucosal defect after polyp removal or not closing the mucosal defect using clips (main intervention and comparison). The resection margins will be approximated using clips. Complete closure is defined as approximated margins with less than 1cm gap between clips. All patients will further be randomized to two different settings of electrocautery (EndoCut or Coagulation) to standardize otherwise variable electrocautery practice, and for explorative analysis.
  Arms: Clip closure + Coagulation; Clip closure + EndoCut

SUMMARY:
The effectiveness of colonoscopy in reducing colorectal cancer mortality relies on the detection and removal of neoplastic polyps. Because the risk of prevalent cancer and of transition to cancer increases with polyp size, effective and safe resection of large polyps is particularly important. Large polyps ≥20mm are removed by so-called endoscopic mucosal resection (EMR) using electrocautery snares. Resection of these large polyps is associated with a risk of severe complications that may require hospitalization and additional interventions. The most common risk is delayed bleeding which is observed in approximately 2-9% of patients. A recent retrospective study suggests that closure of the large mucosal defect after resection may decrease the risk of delayed bleeding. However, significant uncertainty remains about the polypectomy techniques to optimizing resection and minimizing risk. Important aspects that may affect risk include clipping of the mucosal defect and electrocautery setting.

DETAILED DESCRIPTION:
Aim 1. The primary aim of the study is to compare the rate of delayed bleeding complications in patients undergoing endoscopic resection of large polyps between:

* A) Closing the mucosal defect after resection (Clip group) and
* B) Not closing the mucosal defect after resection (No clip group).

Aim 2. The secondary aim of the study is to compare the rate of overall complications in patients undergoing endoscopic resection of large polyps between two cautery settings:

* A) Low power coagulation and
* B) Endocut.

ELIGIBILITY:
Inclusion Criteria:

* Any patient ≥18 and ≤89 who presents for a colonoscopy and who does not have criteria for exclusion
* Patients with a ≥20mm non-pedunculated colon polyp

Exclusion Criteria:

* Patients with known (biopsy proven) invasive carcinoma in a potential study polyp
* Pedunculated polyps (as defined by Paris Classification type Ip or Isp)
* Patients with ulcerated depressed lesions (as defined by Paris Classification type III)
* Patients with inflammatory bowel disease
* Patients who are receiving an emergency colonoscopy
* Poor general health (ASA class>3)
* Patients with coagulopathy with an elevated INR ≥1.5, or platelets <50
* Poor bowel preparation
* Pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 928 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2022-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Pohl, Study Chair — White River Junction VAMC, Geisel School of Medicine at Dartmouth
Locations (1):
- White River Junction VAMC, White River Junction, Vermont, United States

REFERENCES:
- [Derived] Crockett SD, Khashab M, Rex DK, Grimm IS, Moyer MT, Rastogi A, Mackenzie TA, Pohl H; Large Polyp Study Group Consortium. Clip Closure Does Not Reduce Risk of Bleeding After Resection of Large Serrated Polyps: Results From a Randomized Trial. Clin Gastroenterol Hepatol. 2022 Aug;20(8):1757-1765.e4. doi: 10.1016/j.cgh.2021.12.036. Epub 2021 Dec 28. PMID 34971811
- [Derived] Pohl H, Grimm IS, Moyer MT, Hasan MK, Pleskow D, Elmunzer BJ, Khashab MA, Sanaei O, Al-Kawas FH, Gordon SR, Mathew A, Levenick JM, Aslanian HR, Antaki F, von Renteln D, Crockett SD, Rastogi A, Gill JA, Law RJ, Elias PA, Pellise M, Mackenzie TA, Rex DK. Effects of Blended (Yellow) vs Forced Coagulation (Blue) Currents on Adverse Events, Complete Resection, or Polyp Recurrence After Polypectomy in a Large Randomized Trial. Gastroenterology. 2020 Jul;159(1):119-128.e2. doi: 10.1053/j.gastro.2020.03.014. Epub 2020 Mar 12. PMID 32173478
- [Derived] Pohl H, Grimm IS, Moyer MT, Hasan MK, Pleskow D, Elmunzer BJ, Khashab MA, Sanaei O, Al-Kawas FH, Gordon SR, Mathew A, Levenick JM, Aslanian HR, Antaki F, von Renteln D, Crockett SD, Rastogi A, Gill JA, Law RJ, Elias PA, Pellise M, Wallace MB, Mackenzie TA, Rex DK. Clip Closure Prevents Bleeding After Endoscopic Resection of Large Colon Polyps in a Randomized Trial. Gastroenterology. 2019 Oct;157(4):977-984.e3. doi: 10.1053/j.gastro.2019.03.019. Epub 2019 Mar 15. PMID 30885778

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some of the inclusion/exclusion criteria, e.g. polyp size, poor bowel preparation, could not be assessed until after the start of the colonoscopy. Therefore, informed consent was obtained and the patient enrolled in the study prior to the procedure. Only when it was determined that the patient was eligible for the study were they then randomized.
Period: Overall Study
Arm/Group | Clip Closure + EndoCut | Clip Closure + Coagulation | No Clip Closure + EndoCut | No Clip Closure + Coagulation
Started | 227 | 231 | 237 | 233
Crossover (The number of patients who did not receive their designated intervention (clip/no clip).) | 31 | 27 | 22 | 25
Completed | 227 | 228 | 234 | 230
Not Completed | 0 | 3 | 3 | 3
Not completed — no 30-day follow-up data | 0 | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clip Closure + EndoCut | Clip Closure + Coagulation | No Clip Closure + EndoCut | No Clip Closure + Coagulation | Total
Number analyzed (Participants) | 227 | 231 | 237 | 233 | 928
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.7) | 65.5 (9.2) | 64.8 (9.8) | 65.3 (9.8) | 65.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 98 | 96 | 90 | 376
  Male | 135 | 133 | 141 | 143 | 552
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 1 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 16 | 18 | 11 | 17 | 62
  White | 200 | 202 | 214 | 205 | 821
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 9 | 11 | 9 | 38
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (6.6) | 29.0 (5.6) | 29.1 (6.2) | 29.1 (5.6) | 29.2 (6.0)
ASA Class [Count of Participants; unit: Participants] — The American Society of Anesthesiologist (ASA) Classification is a grading system to assess a patient's fitness before undergoing a surgical procedure.
  Participants
    ASA I - normal healthy patient | 23 | 17 | 19 | 20 | 79
    ASA II - patient with mild systemic disease | 125 | 133 | 134 | 121 | 513
    ASA III - patient with severe systemic disease | 79 | 81 | 84 | 92 | 336
Periprocedural Antithrombic Medications [Count of Participants; unit: Participants]
  Antiplatelet agents | 54 | 47 | 61 | 70 | 232
  Anticoagulants | 5 | 15 | 13 | 16 | 49
  None | 168 | 169 | 163 | 147 | 647
Procedure Sedation [Count of Participants; unit: Participants]
  No Sedation | 1 | 4 | 0 | 1 | 6
  Moderate Sedation | 32 | 26 | 33 | 25 | 116
  Monitored Anesthesia | 194 | 201 | 204 | 207 | 806
Quality of Bowel Preparation [Count of Participants; unit: Participants]
  Excellent | 62 | 64 | 55 | 68 | 249
  Good | 123 | 133 | 146 | 127 | 529
  Fair | 42 | 34 | 36 | 38 | 150
Electrocautery [Count of Participants; unit: Participants]
  Forced Coagulation | 0 | 228 | 0 | 230 | 458
  EndoCut | 227 | 0 | 234 | 0 | 461
  None - did not complete study | 0 | 3 | 3 | 3 | 9
Additional Polyps (any size) [Count of Participants; unit: Participants]
  Yes | 98 | 103 | 103 | 104 | 408
  No | 129 | 128 | 134 | 129 | 520
More Than One Study Polyp [Count of Participants; unit: Participants]
  Yes | 19 | 10 | 21 | 11 | 61
  No | 208 | 221 | 216 | 222 | 867

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Delayed Bleeding Complications
Description: A bleeding event that occurred within 30 days after completion of the colonoscopy with a study polyp resection and is associated with a decrease in hemoglobin by at least 2gm, hemodynamic instability, presentation to the ED, need for hospitalization, repeat colonoscopy, or other interventions.
Time Frame: 30 days following a study polyp resection
Population: As per study protocol, the primary analysis was done using clip/no clip closure as the study groups. Data for 9 patients was not available.
Measure: Count of Participants; unit: Participants
Groups:
- Clip Closure: Clipping of the mucosal defect after resection of a ≥20mm non-pedunculated study polyp using clips. Resection is done using the EndoCut electrocautery mode or the Coagulation electrocautery mode.
  Clip closure: Patients will be randomized to either closing the mucosal defect after polyp removal or not closing the mucosal defect using clips (main intervention and comparison). The resection margins will be approximated using clips. Complete closure is defined as approximated margins with less than 1cm gap between clips. All patients will further be randomized to two different settings of electrocautery (EndoCut or Coagulation) to standardize otherwise variable electrocautery practice, and for explorative analysis.
- No Clip Closure: No clipping of the mucosal defect after resection of a ≥20mm non-pedunculated study polyp. Resection is done using the EndoCut electrocautery mode or the Coagulation electrocautery mode.
Arm/Group | Clip Closure | No Clip Closure
Number analyzed (Participants) | 455 | 464
Participants | 16 | 33

2. Secondary Outcome: The Overall Number of Complications
Description: Overall complications are defined as an aggregate of all complications that occur at the time of the procedure (immediate complications) or during 30 days of follow-up. They include delayed bleeding complications, perforation, postpolypectomy syndrome, and clinical events that require an ED visit, admission to the hospital, additional testing or an intervention.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clip Closure | No Clip Closure
Number analyzed (Participants) | 455 | 464
Participants | 22 | 44

3. Secondary Outcome: Complete Study Polyp Resection Rate
Description: Rate of complete study polyp resection at the initial colonoscopy and at first follow-up endoscopy
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Polyp Recurrence Rate
Description: Rate of recurrent polyp at the resection site after complete polyp resection.
Time Frame: 3 months to 5 years
Reporting Status: Not Posted

5. Secondary Outcome: The Number of Complications Associated With Clip Use
Description: Incidence of complications associated with application of clips.
Time Frame: 30 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Measured Factors Associated With Resection Complications
Description: Factors that may be associated with complications, including electrocautery setting, polyp size, location of the polyp in the colon (right, left, rectum), histology, polyp morphology, time required for resection.
Time Frame: 30 days
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Measured Factors Associated With Incomplete Resection or Recurrence of Polyps
Description: Factors that may be associated with incomplete resection may include prior attempts of removal, use of adjunctive argon plasma coagulation for residual polyp removal, polyp size, location, histology.
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Within 30 days of the colonoscopy.
Description: Patients who crossed over (i.e. in the control group, but underwent clip closure) are analyzed as intention to treat, and are therefore analyzed in the control group. Therefore the number of patients at risk equals the number of patients in each group with available follow-up data. For non-SAEs, the number affected does not equal to the number of events because some patients reported multiple adverse events.
Arm/Group | Clip Closure + EndoCut | Clip Closure + Coagulation | No Clip Closure + EndoCut | No Clip Closure + Coagulation
All-Cause Mortality (participants affected / at risk) | 0/227 | 0/228 | 2/234 | 0/230
Serious Adverse Events (participants affected / at risk) | 11/227 | 11/228 | 21/234 | 23/230
Other Adverse Events (participants affected / at risk) | 34/227 | 20/228 | 33/234 | 21/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clip Closure + EndoCut (N=227) | Clip Closure + Coagulation (N=228) | No Clip Closure + EndoCut (N=234) | No Clip Closure + Coagulation (N=230)
Postprocedure hemorrhage (Surgical and medical procedures) | 6 | 10 | 16 | 17
Intraprocedural bleeding (Surgical and medical procedures) | 1 | 0 | 0 | 0
Abdominal Pain (Surgical and medical procedures) | 0 | 1 | 1 | 1
Perforation (Surgical and medical procedures) | 3 | 0 | 3 | 3
Postpolypectomy syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Other (General disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clip Closure + EndoCut (N=227) | Clip Closure + Coagulation (N=228) | No Clip Closure + EndoCut (N=234) | No Clip Closure + Coagulation (N=230)
Abdominal Pain (Gastrointestinal disorders) | 11 (11) | 10 (10) | 11 (11) | 7 (7) — Does not include abdominal pain caused by perforation nor post-polypectomy syndrome.
Bleeding (Gastrointestinal disorders) | 15 (15) | 5 (5) | 16 (16) | 16 (16) — Post procedure bleeding.
Blood pressure problems (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Reports of either hypo or hypertension following the procedure.
Bowel movement problems (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2) — Either constipation or diarrhea following the colonoscopy.
Urinary issues (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) — Reports of urinary tract infection following the procedure.
Cardiovascular event (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headaches/Fevers (General disorders) | 1 (1) | 4 (4) | 3 (3) | 1 (1)
Other (General disorders) | 6 (6) | 5 (5) | 3 (3) | 2 (2) — Used when only a few cases were reported. This category includes fatigue, rash, vomiting, feeling sore, eye pain, possible allergic reaction or cramps.
Post-polypectomy syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Complete defect closure not possible in 13% of patients. Crossover to clip group in 10% of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT01936948/Prot_SAP_000.pdf